CLINICAL TRIAL: NCT07065175
Title: KANGFUPEN (Liquid Dressing) for the Treatment of Chronic Radiation-Induced Rectal Injury: A Prospective, Single-Arm, Multicenter Study
Brief Title: KANGFUPEN Liquid Dressing for Chronic Radiation-Induced Rectal Injury
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University First Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Beijing Rectum Hospital (Unknown); Jilin City Hospital of Chemical Industry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHKANGFUPENG
Record Dates: First submitted 2025-05-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Radiation-induced Proctitis
Keywords: Radiotherapy complications; Chronic radiation-induced proctitis

STUDY DESIGN:
Intervention Model Description: The efficacy assessment employs a repeated-measures design with intra-individual comparisons between baseline and post-treatment timepoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All enrolled patients (Experimental): All enrolled patients receive the same investigational intervention (Kangfupen liquid dressing enema). Scientific comparison is achieved through Pre- vs. post-treatment (3/6/12mo) parameter changes (e.g., ΔLENT-SOMA).
  Interventions: Drug: Kangfupen (liquid dressing) retention enema administration

INTERVENTIONS:
Drug: Kangfupen (liquid dressing) retention enema administration — Dosage: 50 mL per administration, once daily Duration: 3-6 months of continuous therapy
  Procedure:
  Enema depth determined by colonoscopy-identified lesion location Administered as retention enema (minimum 30-minute retention time)

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of Kangfupen (a topical liquid dressing) in treating chronic radiation-induced proctitis (RTOG Grade 2 or higher). The key questions we aim to answer are:

1. Does Kangfupen improve LENT-SOMA rectal injury scores after 3 months of treatment?
2. Does Kangfupen reduce endoscopic inflammation (Vienna score) and symptoms (RTOG/CTCAE grades)?
3. What adverse events occur with Kangfupen therapy? Kangfupen liquid dressing (50 mL/once daily) will be administered as retention enema for 3-6 months, adjusted based on lesion location.

Researchers will evaluate the following outcomes to assess Kangfupen's efficacy and safety in treating chronic radiation proctitis:

1. Change in LENT-SOMA rectal injury score (baseline vs. 3 months).
2. Changes in Vienna endoscopic score, RTOG/CTCAE grades, and IBDQ quality-of-life scores.
3. Symptom improvement rate and time to complete remission.

Participant will:

1. Undergo baseline and 3-month endoscopic evaluations.
2. Complete symptom diaries and quality-of-life questionnaires.
3. Attend regular clinic visits for safety monitoring.

DETAILED DESCRIPTION:
Baseline Assessments

All enrolled patients must complete the following evaluations:

1. Medical history including primary tumor type, histopathology, staging and radiotherapy details (timing, technique, and total dose)
2. Physical examination
3. ECOG performance status
4. Laboratory tests including complete blood count, stool occult blood, liver/kidney function and tumor markers
5. Pelvic scans to exclude tumor recurrence/progression
6. Full colonoscopy with photographic documentation. Images every 5cm from anus to splenic flexure, and at sites of severe mucosal reaction additionally
7. Grading based on LENT-SOMA, RTOG, and CTCAE v5.0 criteria

Treatment protocol Kangfupen (liquid dressing) retention enema

* Dosage: 50 mL once daily for 3-6 months
* Administration depth: Determined by colonoscopy findings Enema preparation & administration 1. Reconstitution:

  1. Transfer liquid from plastic to brown glass vial
  2. Shake vigorously to dissolve lyophilized powder
  3. Return solution to plastic bottle and shake again 2. Delivery:

  <!-- -->

  1. Position: Left lateral decubitus with waste basin
  2. Slowly instill 50 mL into rectum
  3. Retain for ≥30 minutes, rotating positions every 15 minutes (left/right lateral, supine, knee-chest)

Concomitant therapies Permitted: probiotics, smectite, antibiotics, stool softeners Prohibited: 5-ASA drugs (mesalazine/sulfasalazine), endoscopic hemostasis (e.g., argon plasma coagulation), formaldehyde/HBO/surgery/fecal microbiota transplant, other enema therapies.

Toxicity monitoring Potential adverse events include allergic reactions and mechanical injury (bleeding/perforation). Required Actions include immediately discontinuing treatment and reporting to the principal investigating site within 24 hours.

All adverse events will be assessed using CTCAE v5.0 criteria.

Follow-up schedule Month 1-2: LENT-SOMA, RTOG/CTCAE grades, IBDQ, symptom improvement evaluation Month 3: Above + sigmoidoscopy with Vienna scoring Every 6 months after month 6: sigmoidoscopy + all scales + physician's global assessment of treatment efficacy

ELIGIBILITY:
Inclusion Criteria:

* Fully voluntary with decision-making capacity
* 18-80 years old
* Completed pelvic radiotherapy for malignancy ≥3 months prior
* Evidence of chronic radiation-induced rectal injury (RTOG Grade ≥2)
* Evidence of radiation-induced rectal injury on colonoscopy (within 3 months, Vienna endoscopic score ≥1)
* No prior surgery
* ECOG score 0-2
* Estimated survival ≥1 year

Exclusion Criteria:

* Primary rectal tumours or pelvic malignancies with rectal involvement
* Uncontrolled, recurrent, or metastatic tumours
* Concurrent anticancer therapies including radiotherapy, chemotherapy, targeted therapy, immunotherapy and traditional Chinese medicine with anti-tumour properties
* Patients with intestinal fistula, perforation, or obstruction
* History of electrocautery treatment within 1 month
* Recent medication use (within 2 weeks): traditional Chinese medicine enemas, mesalazine (oral or rectal) and other anti-inflammatory bowel medications
* History of superoxide dismutase allergy
* Pre-existing chronic colitis, ulcerative colitis, or nonspecific proctitis
* Connective tissue diseases requiring long-term corticosteroid therapy
* Pregnant or lactating women
* Active infection or fever
* Other severe comorbidities potentially affecting trial compliance: unstable cardiac disease requiring treatment, renal disorders, chronic hepatitis, poorly controlled diabetes and psychiatric illnesses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in LENT-SOMA rectal radiation injury scores from baseline to 3 months post-treatment | From enrolment to 3 months post-treatment
  Treatment response is defined as:
  1. Effective: Decrease in LENT-SOMA score compared to baseline
  2. Ineffective: No change or increase in LENT-SOMA score versus baseline

SECONDARY OUTCOMES:
Change in Vienna endoscopic scores from baseline to post-treatment | From enrolment to 3 months post-treatment
  Treatment response is defined as:
  1. Effective: Any decrease in Vienna endoscopic score at 3 months post-treatment compared to baseline
  2. Ineffective: Stable or increased score compared to baseline
Changes in RTOG and CTCAE grading from baseline to post-treatment assessments | From enrolment to 3 months post-treatment
  Treatment response is defined as:
  1. Efficient: Any decrease in either RTOG radiation toxicity grade or CTCAE adverse event grade from baseline
  2. Inefficient: No improvement or worsening in both grading systems
Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Function and Bleeding Scores from baseline to post-treatment | From enrolment to 3 months post-treatment
  Treatment response is defined as:
  1. Efficient: Any decrease in IBDQ bowel function and bleeding scores post-treatment compared to baseline
  2. Inefficient: No change or increase in IBDQ bowel function and bleeding scores versus baseline
Post-treatment symptom improvement rate | From enrolment to 3 months post-treatment
  Symptoms are categorized into:
  Complete remission: Complete resolution of clinical symptoms (e.g., rectal bleeding, diarrhea, tenesmus) Partial remission: Significant improvement in symptoms, but not complete resolution Stable disease: No significant change in symptoms (no improvement or worsening) Progression: Worsening of clinical symptoms
  Treatment response is defined as:
  1. Effective: Complete remission or partial remission
  2. Ineffective: Stable disease or progression

OTHER OUTCOMES:
Endoscopic response (Vienna Score) | From enrolment to 6, 12, 24, 36 months post-treatment
  Assessment: Change from baseline at each timepoint
  Response Criteria:
  Effective: Decreased Vienna score Ineffective: Stable/increased score
Toxicity improvement (RTOG/CTCAE) | From enrolment to 6, 12, 24, 36 months post-treatment
  Assessment: Grading change from baseline
  Response Criteria:
  Effective: Reduced RTOG/CTCAE grade Ineffective: Unchanged/worsened grade
Quality of life (IBDQ Bowel Function/Bleeding) | From enrolment to 6, 12, 24, 36 months post-treatment
  Assessment: Subscore change from baseline
  Response Criteria:
  Effective: Score reduction (symptom improvement) Ineffective: Stable/elevated score
Symptom improvement rate | From enrolment to 6, 12, 24, 36 months post-treatment
  Categories:
  Complete Response (CR): Total symptom resolution (RTOG Grade 0) Partial Response (PR): ≥50% symptom reduction Stable Disease (SD): No significant change Progression (PD): Symptom worsening Clinical Benefit: CR + PR Note: For discordant symptoms, the primary symptom (investigator-designated) determines classification.
Time to complete symptom resolution | From enrolment to sustained (≥7 days) CR

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zhu J, Li X, Huang M, Zhu H, Tan Y, He X, Sun Z, Cheng H, Li F, Jiang P, Lou H, Ke G, Cao X, Zhu L, Xie P, Yan J, Zhang F. Application of Recombinant Human Superoxide Dismutase in Radical Concurrent Chemoradiotherapy for Cervical Cancer to Prevent and Treat Radiation-induced Acute Rectal Injury: A Multicenter, Randomized, Open-label, Prospective Trial. Int J Radiat Oncol Biol Phys. 2024 Nov 1;120(3):720-729. doi: 10.1016/j.ijrobp.2024.04.070. Epub 2024 May 4. PMID 38705489
- [Background] Tohidinezhad F, Willems Y, Berbee M, Limbergen EV, Verhaegen F, Dekker A, Traverso A. Prediction models for brachytherapy-induced rectal toxicity in patients with locally advanced pelvic cancers: a systematic review. J Contemp Brachytherapy. 2022 Aug;14(4):411-422. doi: 10.5114/jcb.2022.119427. Epub 2022 Aug 31. PMID 36199943
- [Background] Michalski JM, Yan Y, Watkins-Bruner D, Bosch WR, Winter K, Galvin JM, Bahary JP, Morton GC, Parliament MB, Sandler HM. Preliminary toxicity analysis of 3-dimensional conformal radiation therapy versus intensity modulated radiation therapy on the high-dose arm of the Radiation Therapy Oncology Group 0126 prostate cancer trial. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):932-8. doi: 10.1016/j.ijrobp.2013.07.041. Epub 2013 Oct 8. PMID 24113055
- [Background] Wang CJ, Huang EY, Sun LM, Chen HC, Fang FM, Hsu HC, Changchien CC, Leung SW. Clinical comparison of two linear-quadratic model-based isoeffect fractionation schemes of high-dose-rate intracavitary brachytherapy for cervical cancer. Int J Radiat Oncol Biol Phys. 2004 May 1;59(1):179-89. doi: 10.1016/j.ijrobp.2003.10.025. PMID 15093915